CLINICAL TRIAL: NCT04658407
Title: Patients' Outcome With Severe or Fulminant Hepatic Insufficiency, Hospitalized in the Hospitals of the Assistance Publique - Hôpitaux de Paris (APHP)
Brief Title: Patients' Outcome With Severe or Fulminant Hepatic Insufficiency, Hospitalized in the Public Hospitals of Paris
Acronym: DEVINHEF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AP-HP200240
Record Dates: First submitted 2020-09-21; First posted 2020-12-08 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2020-09

CONDITIONS: Fulminating Hepatic Failure
MeSH Terms: conditions — Liver Failure, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- all patients diagnosed with a severe hepatic failure: Retrospective cohort using only data already entered in the Health data warehouse of the APHP (Public Paris Hospital)

SUMMARY:
The main objective is to determine the medical fate (transplanted or not and living or deceased), of patients with Severe, fulminating acute liver failure in the public hospitals of paris.

DETAILED DESCRIPTION:
Severe, fulminating acute liver failure is a rare but serious disease. The overall prognosis has improved in recent years thanks to advances in medical management and liver transplantation.

However, the epidemiology of this disease in France, the survival with or without liver transplantation of these patients and the factors that can influence this survival are not well known.

The main objective is to determine the medical fate (transplanted or not and living or deceased), of patients with Severe, fulminating acute liver failure in the public hospitals of paris (APHP).

The data will come from the APHP Health Data Warehouse

ELIGIBILITY:
Inclusion Criteria:

* Age > 15
* Severe liver failure or toxicants that may cause a liver failure Or
* (PR<50% or INR >1.5) And ALT >250

Exclusion Criteria:

* Patients with underlying chronic liver disease
* Patients with the conditions given by this following ICD (International Classification of Diseases) : B18 - E831 - K70 - K715 - K717 - K730- K731 - K732 - 738 - K74 - K753 - K758 - K760 - K761

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with Severe liver failure or toxicants that may cause a liver failure
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
The main objective is to determine the medical fate (transplanted or not and living or deceased), of patients with Severe and fulminating acute hepatic failure within AP-HP hospitals | 1 month from the diagnosis of this episode
  Patient status 1 month after diagnosis of this episode (alive or dead with or without transplantation)

SECONDARY OUTCOMES:
Epidemiology of Severe and fulminating acute hepatic failure | Baseline
  Sex Ratio M / F and cause of liver failure
Cause of death | From date of inclusion until the date of death from any cause, assessed up to 9 years
  Cause of death
Analysis of Clinical Pathway | up to 1month after the diagnosis of this episode
  Identification of the different services visited
Reasons for new hospitalizations with an admission date within 6 months after the diagnosis this episode | within 6 months after the diagnosis this episode
  Identification by the usual code of the new hospitalization, consecutive to the episode

CONTACTS AND LOCATIONS:
Locations (1):
- Paul Brousse Hospital, Villejuif, France

IPD SHARING:
Plan to Share IPD: No